CLINICAL TRIAL: NCT05069792
Title: Utrecht COhort for Lung Cancer Outcome Reporting and Trial Inclusion (U-COLOR)
Acronym: U-COLOR
Status: Active, not recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Professor, UMC Utrecht
Other Study IDs: NL71047.041.19
Record Dates: First submitted 2021-09-09; First posted 2021-10-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Objective: 1) To collect information on patient characteristics, short- and long-term clinical and patient-reported outcomes; and 2) to create an infrastructure for efficient, fast, and pragmatic randomized evaluation of new interventions.

Study design: Observational, prospective cohort study, according to the 'TwiCs' design.

Study population: All patients with lung cancer referred to the Department of Pulmonology or the Department of Radiotherapy of the UMC Utrecht.

Main study parameters/endpoints: Clinical parameters (performance status, co-morbidity, oncological history, symptoms, imaging, technical and treatment data), clinical endpoints (toxicity, reintervention and survival), and patient-reported outcomes.

DETAILED DESCRIPTION:
The prospective U-COLOR cohort (Utrecht COhort for Lung cancer Outcome Reporting and trial inclusion), aims to:

* Gather data on natural disease progression, treatment response, disease recurrence, complications, quality of life and survival of patients with lung cancer;
* Collect a patient group willing to participate in studies;
* Facilitate multiple, parallel randomized controlled trials within the cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Radiographic and/or histologic proof of lung cancer;
* Referred to Department of Pulmonology or the Department of Radiotherapy for treatment.

Exclusion Criteria:

* Mental disorder or cognitive dysfunction that hinders the patient's ability to understand the informed consent procedure and/or study details;
* Patients with severe psychiatric disorders;
* Inability to understand the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are referred to the Department of Pulmonology or the Department of Radiotherapy of the UMC Utrecht for treatment of lung cancer will be eligible to be enrolled in the U-COLOR cohort.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Change in Health-related Quality of Life | Up to 10 years after treatment
  Assesment of Health-related quality of life in lung cancer patients undergoing treatment
Occurence of toxicity (adverse events) | Up to 10 years after treatment
  Grade ≥3 side effects occurring during or up to 3 months after radiotherapy will be registered according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0). For 'dysphagia' and 'pneumonitis' endpoints, also grade 2 toxicity will be scored.
Readmission | Up to 10 years after treatment
  Reintervention (re-irradiation, surgery, other), tube feeding requirement or treatment for local and/or distant progression.
Survival | Up to 10 years after treatment
  Date of last follow-up, date of local progression, date of distant progression, location of distant progression. Overall survival (Survival of participating patients will be recorded using the follow up questionnaires [returned by family members] or are derived from the Statistic Netherlands Database [in Dutch: Centraal Bureau voor de Statistiek, CBS] and Dutch Cancer Registry [in Dutch: Integraal Kankercentrum Nederland, IKNL]).

CONTACTS AND LOCATIONS:
Overall Officials: Helena M Verkooijen, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands